CLINICAL TRIAL: NCT06429774
Title: Comparative Effectiveness of Intervention in Multi-level Hospitals for Acute Traumatic Brain Injury: a Prospective, Multicenter, Observational Cohort Study
Brief Title: Comparative Effectiveness of Intervention in Multi-level Hospitals for Acute Traumatic Brain Injury(Metric-TBI)
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Weiming Liu, Professor, Beijing Tiantan Hospital
Other Study IDs: SF 2024-1-2042
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Beijing-Tianjin-Hebei region; Database; Comparative effectiveness of intervention; Clinical Treatment Guideline
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Nervous System Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — * vein blood
  * hematoma fluid
  * dura mater
  * hematoma outer membrane
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TBI Group: TBI patients recruited from neurosurgical departments at 50 medical centers in China have apparent clinical symptoms that are confirmed by computed tomography or magnetic resonance imaging.
  The exclusion criteria are those who fulfill one of the following conditions:
  1. patients ≥90 years of age;
  2. patients who did not accept follow-up visits or were unable to complete follow-up assessments;
  3. patients with incomplete information;
  4. patients who did not obtain written informed consent;
  5. patients with concomitant cancer or other serious illnesses.
  Interventions: Other: Neurological function; Other: Mental State, cognitive function, and life quality assessment; Other: Peripheral blood test; Other: Hematoma test

INTERVENTIONS:
Other: Neurological function — Neurological function will be examined using Glasgow Coma Scale (GCS) and Extended Glasgow Outcome Scale (GOSE).The GOSE was created as an advancement from the original GOS. The GOSE score categorizes the prognosis of patients with traumatic brain injury into eight categories.The 8 categories are: Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper Moderate Disability, Lower Good Recovery, and Upper Good Recovery.
Other: Mental State, cognitive function, and life quality assessment — Mental State, cognitive function, and life quality will be examined using the Generalized Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9(PHQ-9), Rivermead post-concussion symptoms questionnaire(RPQ), PTSD Checklist-5 Version(PCL-5)，Six-Item Screener（SIS） and 12-Item Short-Form Health Survey version 2(SF-12v2).
Other: Peripheral blood test — Collect peripheral blood samples from patients.
Other: Hematoma test — Collect hematoma fluid, dura mater, and hematoma outer membrane samples from patients.

SUMMARY:
A prospective, multicenter, observational cohort study is designed to compare the effectiveness of intervention in multi-grade hospitals for acute traumatic brain injury and to optimize clinical outcomes.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is associated with significant morbidity, mortality, and disability, profoundly impacting public health. This study aims to establish a database for acute craniocerebral trauma within the Beijing-Tianjin-Hebei region, and compiles indicators of hospital treatment capabilities and patient data, including neuroimaging, clinical progression, and rehabilitation prognoses.The study is bifurcated into two segments: the initial phase surveys the current status of acute treatment outcomes for TBI inpatients across hospitals in the Beijing-Tianjin-Hebei region and conducts a comparative effectiveness analysis to identify the clinical interventions to optimize. Subsequent phases build on the former by applying optimized treatment strategies to improve efficacy and establish collaborative optimized treatment protocols.

This is a prospective, multicenter, observational study designed to enroll 2,000 patients under the age of 90 years with traumatic brain injury in the presence of clinical symptoms confirmed by computed tomography or magnetic resonance imaging.The primary outcome is the Extended Glasgow Outcome Score within 12 months. Secondary outcomes include the Generalized Anxiety Disorder-7 (GAD-7), Patient Health Questionnaire-9(PHQ-9), Rivermead post-concussion symptoms questionnaire(RPQ), PTSD Checklist-5 Version(PCL-5)，Six-Item Screener (SIS) and 12-Item Short-Form Health Survey version 2(SF-12v2).

The objective of this study is anticipated to the Beijing-Tianjin-Hebei region a 20 percent increase in the number of cases treated by optimized clinical practice guidelines and a 10 percent decrement in mortality and disability rates among TBI patients in the region.

ELIGIBILITY:
Inclusion Criteria:

* Patient (1 years to 89 years) presenting with clinical symptoms of traumatic brain injury
* Traumatic brain injury verified on cranial computed tomography or magnetic resonance imaging
* Written informed consent from patients or their next of kin according to the patient's cognitive status

Exclusion Criteria:

* patients ≥90 years of age
* patients who did not accept follow-up visits or were unable to complete follow-up assessments
* patients with incomplete information
* patients who did not obtain written informed consent
* patients with concomitant cancer or other serious illnesses

Ages: 1 Year to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: TBI patients recruited from neurosurgical departments at 50 medical centers in China have apparent clinical symptoms that are confirmed by computed tomography or magnetic resonance imaging.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the Extended Glasgow Outcome Score | From discharge up to 12 months postoperatively
  The Extended Glasgow Outcome Scores(GOSE) range from 1 to 8, with higher scores indicating a better outcome. The summary of the scale is below:1.Dead;2. Vegetative State;3. Lower Severe Disability;4. Upper Severe Disability;5. Lower Moderate Disability;6. Upper Moderate Disability;7. Lower Good Recovery;8.Upper Good Recovery.Therefore, a score of 1 represents the worst outcome (death), and a score of 8 represents the best outcome (upper good recovery).
  The rates of death or severe disability (GOSE scores 1-3) due to traumatic brain injury in the short term (at discharge) and in the long term (3, 6, and 12 months post-discharge) give an indication of the extent to which a patient recovers from different treatments.

SECONDARY OUTCOMES:
Difference in the Generalized Anxiety Disorder-7 Scale in post-traumatic mental health recovery | From discharge up to 12 months postoperatively
  Patients were scored on their subsequent level of mental health at 3, 6, and 12 months after discharge based on the Generalized Anxiety Disorder-7 Scale(GAD-7).
  The GAD-7 scale consists of seven items, each describing a symptom of Generalized Anxiety Disorder(GAD), and respondents rate how often they've been bothered by each symptom over the past two weeks.The GAD-7 score of 10 suggests moderate anxiety, on a scale ranging from 0 (minimal anxiety) to 21 (severe anxiety), with higher scores indicating worse outcomes.
Difference in the Patient Health Questionnaire-9 Scale in post-traumatic mental health recovery | From discharge up to 12 months postoperatively
  Patients were scored on their subsequent level of mental health at 3, 6, and 12 months after discharge based on the Patient Health Questionnaire-9 Scale(PHQ-9).
  The PHQ-9 scale consists of nine items, each describing a symptom of depression, and respondents rate how often they've been bothered by each symptom over the past two weeks. The PHQ-9 scores between 10-14 suggest moderate depression, on a scale ranging from 0 (minimal depression) to 27 (severe depression), with higher scores indicating worse outcomes.
Difference in the Rivermead Post-Concussive Symptoms Questionnaire Scale in post-traumatic mental health recovery | From discharge up to 12 months postoperatively
  Patients were scored on their subsequent level of mental health at 3, 6, and 12 months after discharge based on the Rivermead Post-Concussive Symptoms Questionnaire(RPQ).
  The RPQ score ranges from 0 (no symptoms) to 64 (severe symptoms). Higher scores on the RPQ indicate a greater severity of post-concussive symptoms and a worse outcome. This information helps healthcare providers assess the impact of the concussion on the patient's daily life and track their recovery progress.
Difference in the Post-Traumatic Stress Disorder Checklist-5 Scale in post-traumatic mental health recovery | From discharge up to 12 months postoperatively
  Patients were scored on their subsequent level of mental health at 3, 6, and 12 months after discharge based on the Post-Traumatic Stress Disorder Checklist-5 (PCL-5). Each of the 20 items on the PCL-5 is rated on a scale from 0 ("Not at all") to 4 ("Extremely"). The PCL-5 score ranges from 0 to 80, with higher scores indicating worse Post-traumatic stress disorder(PTSD) symptoms.
Difference in life quality assessment | From discharge up to 12 months postoperatively
  Patients were scored on their subsequent level of quality of life at 3, 6, and 12 months after discharge based on different scores on the 12-item Short-Form Health Survey 2 (SF-12v2).
  The SF-12v2 provides two summary scores: the Physical Component Summary (PCS) score and the Mental Component Summary (MCS) score. For both the PCS and MCS scores range from 0(the lowest level of health) to 100(the highest level of health). Higher scores on the PCS and MCS indicate better physical and mental health, respectively.
Difference in cognitive function | From discharge up to 12 months postoperatively
  Patients were scored on their subsequent level of cognitive function at 3, 6, and 12 months after discharge based on different scores on the Six-Item Screener (SIS).
  The SIS is a brief cognitive assessment tool used primarily to screen for cognitive impairment. The SIS assesses orientation and recall, two critical components often affected in cognitive disorders such as dementia.It ranges from 0 to 6, with higher scores mean a better outcome in terms of cognitive function.
Rate of complications and adverse events | From discharge up to 12 months postoperatively
  Rates of complications and adverse events during hospitalization and 12 months after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Weiming Liu, M.D., Principal Investigator — Beijing Tiantan Hospital
Locations (64):
- China (64):
  - Beijing Fengtai You'anmen Hospital, Beijing, Beijing Municipality
  - Beijing Huairou Hospital, Beijing, Beijing Municipality
  - Beijing Luhe Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Red Cross Emergency Medical Center, Beijing, Beijing Municipality
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Chaoyang Integrative Medicine Rescue And First Aid Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Changping Hospital, Beijing, Beijing Municipality
  - Beijing Mentougou District Hospital, Beijing, Beijing Municipality
  - Liangxiang Hospital, Beijing, Beijing Municipality
  - The First Hospital of Fangshan District, Bejing, Beijing, Beijing Municipality
  - Dongfang Hospital of Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Affiliated Hospital Of Hebei University, Baoding, Hebei
  - The No.2 Hospital of Baoding, Baoding, Hebei
  - Anguo Hospital, Baoding, Hebei
  - Rongcheng People's Hospital, Baoding, Hebei
  - Xiongxian Hospital, Baoding, Hebei
  - Baoding Seventh Hospital, Baoding, Hebei
  - Gaobeidian Hospital, Baoding, Hebei
  - Yixian Hospital, Baoding, Hebei
  - Suning Hospital, Cangzhou, Hebei
  - Pingquan Hospital, Chengde, Hebei
  - Luanping Hospital, Chengde, Hebei
  - Hangang Hospital, Handan, Hebei
  - Weixian Chinese Traditional Medicine Hospital, Handan, Hebei
  - The No.1 Hospital Of Yongnian District Handan City, Handan, Hebei
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Langfang People's Hospital, Langfang, Hebei
  - Edelburg Hospital, Langfang, Hebei
  - Sanhe Hospital, Langfang, Hebei
  - Yanjiao Fuhe No.1 Hospital, Langfang, Hebei
  - Dachang Hui Autonomous County People's Hospital, Langfang, Hebei
  - Xianghe Hospital, Langfang, Hebei
  - Fourth people's Hospital of Langfang, Langfang, Hebei
  - Dacheng Hospital, Langfang, Hebei
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Shanhaiguan People's Hospital, Qinhuangdao, Hebei
  - Qinhuangdao Funing District Hospital of Traditional Chinese Medicine, Qinhuangdao, Hebei
  - Lulong Hospital, Qinhuangdao, Hebei
  - Peking University Third Hospital Qinhuangdao Hospital, Qinhuangdao, Hebei
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Hospital Of Shijiazhuang, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Jingxing Hospital, Shijiazhuang, Hebei
  - Xinle Chinese Traditional Medicine Hospital, Shijiazhuang, Hebei
  - Tangshan Fengrun People's Hospital, Tangshan, Hebei
  - Tangshan Workers' Hospital, Tangshan, Hebei
  - Xingtai Central Hospital, Xingtai, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Xingtai Xindu District People's Hospital, Xingtai, Hebei
  - Xingtai Nanhe District People's Hospital, Xingtai, Hebei
  - Pingxiang People's Hospital, Xingtai, Hebei
  - Wei County People's Hospital, Xingtai, Hebei
  - Qinghe Central Hospital, Xingtai, Hebei
  - Xingtai Ninth Hospital, Xingtai, Hebei
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Hospital, Tianjin, Tianjin Municipality
  - Tianjin Fourth Central Hospital, Tianjin, Tianjin Municipality
  - Tianjin Xiqing Hospital, Tianjin, Tianjin Municipality
  - Wuqing People's Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capizzi A, Woo J, Verduzco-Gutierrez M. Traumatic Brain Injury: An Overview of Epidemiology, Pathophysiology, and Medical Management. Med Clin North Am. 2020 Mar;104(2):213-238. doi: 10.1016/j.mcna.2019.11.001. PMID 32035565
- [Background] Galgano M, Toshkezi G, Qiu X, Russell T, Chin L, Zhao LR. Traumatic Brain Injury: Current Treatment Strategies and Future Endeavors. Cell Transplant. 2017 Jul;26(7):1118-1130. doi: 10.1177/0963689717714102. PMID 28933211
- [Background] Jiang JY, Gao GY, Feng JF, Mao Q, Chen LG, Yang XF, Liu JF, Wang YH, Qiu BH, Huang XJ. Traumatic brain injury in China. Lancet Neurol. 2019 Mar;18(3):286-295. doi: 10.1016/S1474-4422(18)30469-1. Epub 2019 Feb 12. PMID 30784557
- [Background] Stocchetti N, Carbonara M, Citerio G, Ercole A, Skrifvars MB, Smielewski P, Zoerle T, Menon DK. Severe traumatic brain injury: targeted management in the intensive care unit. Lancet Neurol. 2017 Jun;16(6):452-464. doi: 10.1016/S1474-4422(17)30118-7. PMID 28504109
- [Background] Steyerberg EW, Wiegers E, Sewalt C, Buki A, Citerio G, De Keyser V, Ercole A, Kunzmann K, Lanyon L, Lecky F, Lingsma H, Manley G, Nelson D, Peul W, Stocchetti N, von Steinbuchel N, Vande Vyvere T, Verheyden J, Wilson L, Maas AIR, Menon DK; CENTER-TBI Participants and Investigators. Case-mix, care pathways, and outcomes in patients with traumatic brain injury in CENTER-TBI: a European prospective, multicentre, longitudinal, cohort study. Lancet Neurol. 2019 Oct;18(10):923-934. doi: 10.1016/S1474-4422(19)30232-7. PMID 31526754
- [Background] Silverberg ND, Duhaime AC, Iaccarino MA. Mild Traumatic Brain Injury in 2019-2020. JAMA. 2020 Jan 14;323(2):177-178. doi: 10.1001/jama.2019.18134. No abstract available. PMID 31816030
- [Background] Sun D, Jiang B, Ru X, Sun H, Fu J, Wu S, Wang L, Wang L, Zhang M, Liu B, Wang W; for the NESS-China investigators. Prevalence and Altered Causes of Traumatic Brain Injury in China: A Nationwide Survey in 2013. Neuroepidemiology. 2020;54(2):106-113. doi: 10.1159/000501911. Epub 2019 Dec 18. PMID 31851999